CLINICAL TRIAL: NCT03801291
Title: Transvaginal Versus Transperineal Repair of Anterior Rectocele: a Randomized Controlled Trial
Brief Title: Transvaginal Versus Transperineal Repair of Rectocele
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: masnoura99
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Rectocele
MeSH Terms: conditions — Rectocele

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transvaginal repair (Active Comparator): Repair of anterior rectocele via the vagina
  Interventions: Procedure: Transvaginal repair
- Transperineal repair (Active Comparator): Repair of anterior rectocele via the perineum
  Interventions: Procedure: Transperineal repair

INTERVENTIONS:
Procedure: Transvaginal repair — Vaginal incision through which plication of the rectovaginal septum is done
  Arms: Transvaginal repair
Procedure: Transperineal repair — Perineal incision through which plication of the rectovaginal septum is done
  Arms: Transperineal repair

SUMMARY:
Patients with anterior rectocele were randomized to undergo either transvaginal or transperineal repair. The primary outcome of the study was improvement in constipation at 6 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients with anterior rectocele

Exclusion Criteria:

* Male patients.
* Combined rectocele with internal rectal prolapse.
* Anismus.
* Associated anorectal condition such as hemorrhoids and anal fissure.
* Pregnancy.
* Unwilling to participate in the trial

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only
Enrollment: 64 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Improvement in constipation | 6 and 12 months after surgery
  decrease in Wexner constipation score by 25%

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Balata M, Elgendy H, Emile SH, Youssef M, Omar W, Khafagy W. Functional Outcome and Sexual-Related Quality of Life After Transperineal Versus Transvaginal Repair of Anterior Rectocele: A Randomized Clinical Trial. Dis Colon Rectum. 2020 Apr;63(4):527-537. doi: 10.1097/DCR.0000000000001595. PMID 31996580